CLINICAL TRIAL: NCT04025606
Title: Paravertebral Block Versus Thoracic Epidural Analgesia in Patients Undergoing Video Assisted Lung Surgery
Brief Title: Paravertebral Block Versus Thoracic Epidural Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017/2424
Record Dates: First submitted 2019-06-12; First posted 2019-07-19 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Lung Cancer; Postoperative Pain
Keywords: Epidural analgesia; Pneumonectomy
MeSH Terms: conditions — Lung Neoplasms; Pain, Postoperative | interventions — Tea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thoracic epidural analgesia (Active Comparator): Standard thoracic epidurals preoperatively at the dag of surgery.
  Interventions: Drug: Thoracic epidural
- Paravertebral block (Experimental): Paravertebral block inserted at the end of the operation by the surgeons
  Interventions: Drug: Paravertebral block

INTERVENTIONS:
Drug: Thoracic epidural — Standard thoracic epidural (needle inserted into the space between the covering of spinal cord and the cord itself) preoperatively. Standard thoracic epidural analgesia mixture (2 mg/ ml bupivacaine, 2 µg/ ml fentanyl and 2 µg/ ml adrenalin) with an infusion of 6-10 ml/hour until day 2 postoperatively. Thereafter reduction by 30 % every four hours.
  Arms: Thoracic epidural analgesia
Drug: Paravertebral block — Paravertebral block containing 5 ml bupivacaine 5 mg/ ml (optionally 10 ml bupivacaine 2,5 mg/ ml). In addition per-oral painkillers (oxycodone and paracetamol) from the day of surgery.
  Arms: Paravertebral block

SUMMARY:
Thoracic epidural analgesia (TEA) is the basic method of analgesia in patients undergoing pulmonary lobectomy. TEA is considered to be a safe and thoroughly investigated method of pain relief that rarely causes serious complications. However, blocking the nerves as they emerge from the spinal column (paravertebral block, PVB) may represent an alternative method with some potential benefits. In this study, TEA and PVB will be compared for patients undergoing pulmonary lobectomy by video assisted thoracoscopic surgery. The aim of the study is to test the hypothesis, that PVB is a time-saving procedure compared with TEA on the day of surgery and that PVB is as efficient in postoperative pain reduction as TEA.

ELIGIBILITY:
Inclusion Criteria:

Patients with lung cancer in stage 1 or 2 who are accepted for VATS-lobectomy

Exclusion Criteria, preoperative:

Patients who do not wish to participate

Patients with:

* suspicion of ingrowth in the thoracic wall.
* marginal lung function.
* kidney failure.
* chronic pains and/ or daily use of opioids.
* cognitive, visual and / or linguistic dysfunction.
* allergies to drugs used in the paravertebral block or the thoracic epidural analgesia.

Exclusion Criteria, Per- and postoperative

* conversion from VATS to thoractomy.
* unsuccessful admission of thoracic epidural analgesia
* unsuccessful admission of paravertebral block
* postoperative respiratory treatment
* postoperative delirium Patients who for various reasons are not able to self-report pain after surgery.

Patients who wish to withdraw from the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Time in minutes total time at the operating ward | 1 hour
Pain intensity during hospitalization: Numerical Rating Scale (NRS) | Up to 12 months after surgery
  using the Numerical Rating Scale (NRS) in predetermined time intervals after the operation

SECONDARY OUTCOMES:
Hospital length of stay in days | until discharge from hospital (max 1 month)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Wahba, md phd, Study Director — St. Olavs Hospital
Locations (1):
- St Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No